CLINICAL TRIAL: NCT01512160
Title: A Randomized, Double-Blind Third Party Open, Double-Dummy, Parallel Group, Placebo Controlled Study Assessing The Efficacy Of Single Doses Of Pf-04531083 For The Treatment Of Post-Surgical Dental Pain Using Ibuprofen 400 Mg As A Positive Control
Brief Title: Efficacy Of Pf-04531083 In Treating Post-Surgical Dental Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B1351010
Record Dates: First submitted 2011-08-30; First posted 2012-01-19 (Estimated); Results first posted 2013-06-28 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-05

CONDITIONS: Post-surgical Dental Pain
Keywords: Post-surgical dental pain
MeSH Terms: interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- PF-04531083 2000 mg (Experimental)
  Interventions: Drug: PF-04531083; Other: Placebo
- PF-04531083 1000 mg (Experimental)
  Interventions: Drug: PF-04531083; Other: Placebo
- Ibuprofen 400 mg (Active Comparator)
  Interventions: Drug: Ibuprofen; Other: Placebo
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PF-04531083 — 2000 mg oral solution
  Arms: PF-04531083 2000 mg
Other: Placebo — Placebo tablets for Ibuprofen
  Arms: PF-04531083 2000 mg
Drug: PF-04531083 — 1000 mg oral solution
  Arms: PF-04531083 1000 mg
Other: Placebo — Placebo tablets for Ibuprofen
  Arms: PF-04531083 1000 mg
Drug: Ibuprofen — 2 x 200 mg tablets
  Arms: Ibuprofen 400 mg
Other: Placebo — Placebo solution for PF-04531083
  Arms: Ibuprofen 400 mg
Other: Placebo — Placebo solution for PF-04531083
  Arms: Placebo
Other: Placebo — Placebo tablets for Ibuprofen
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the overall pain relief of a single dose of PF-04531083 against placebo following third molar extraction.

ELIGIBILITY:
Inclusion Criteria:

* Oral surgical procedure having removed 2 third molars (unilateral).
* Pre-dose pain intensity score (100 mm Visual Analog Scale [VAS]) >50 mm within 5 hours of oral surgery.
* Pre-dose pain intensity score of moderate or within 5 hours of oral surgery.

Exclusion Criteria:

* Presence or history of any significant hepatic, renal, endocrine, cardiovascular, neurological (including subjects with a history of frequent moderate to severe headaches or subjects with episodic migraines more than twice per month), psychiatric, gastrointestinal, pulmonary, hematologic, or metabolic disorder.
* Prior use of any type of analgesic or NSAID within five half-lives of that drug or less before taking the first dose of study medication, except for anesthesia for the procedure.
* Recent history of chronic analgesic or tranquilizer dependency.
* Active dental infection at the time of surgery.
* Any significant oral surgery complication at the time of surgery or in the immediate postoperative period or dental surgery lasting > 30 minutes.
* Subjects who are smokers.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2011-10; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Austin, Texas, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1351010&StudyName=Efficacy%20Of%20Pf-04531083%20In%20Treating%20Post-Surgical%20Dental%20Pain

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-04531083 1000 mg: Single oral dose of PF-04531083 1000 milligram (mg) spray dried dispersion presented as an oral solution along with 2 placebo tablets matched to ibuprofen 200 mg (equivalent to ibuprofen 400 mg) 1 to 5 hours post-surgery in participants with post-surgical pain intensity of moderate to severe, and confirmed by a score of at least 50 millimeter (mm) on a 100 mm Visual Analogue Scale (VAS).
- PF-04531083 2000 mg: Single oral dose of PF-04531083 2000 mg spray dried dispersion presented as an oral solution along with 2 placebo tablets matched to ibuprofen 200 mg (equivalent to ibuprofen 400 mg) 1 to 5 hours post-surgery in participants with post-surgical pain intensity of moderate to severe, and confirmed by a score of at least 50 mm on a 100 mm VAS.
- Ibuprofen 400 mg: Single oral dose of 2 ibuprofen 200 mg tablets (equivalent to ibuprofen 400 mg) along with placebo matched to PF-04531083 spray dried dispersion presented as an oral solution 1 to 5 hours post-surgery in participants with post-surgical pain intensity of moderate to severe, and confirmed by a score of at least 50 mm on a 100 mm VAS.
- Placebo: Single oral dose of placebo matched to PF-04531083 spray dried dispersion presented as an oral solution along with 2 placebo tablets matched to ibuprofen 200 mg (equivalent to ibuprofen 400 mg) 1 to 5 hours post-surgery in participants with post-surgical pain intensity of moderate to severe, and confirmed by a score of at least 50 mm on a 100 mm VAS.
Period: Overall Study
Arm/Group | PF-04531083 1000 mg | PF-04531083 2000 mg | Ibuprofen 400 mg | Placebo
Started | 22 | 23 | 22 | 23
Completed | 20 | 23 | 22 | 22
Not Completed | 2 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- PF-04531083 1000 mg: Single oral dose of PF-04531083 1000 mg spray dried dispersion presented as an oral solution along with 2 placebo tablets matched to ibuprofen 200 mg (equivalent to ibuprofen 400 mg) 1 to 5 hours post-surgery in participants with post-surgical pain intensity of moderate to severe, and confirmed by a score of at least 50 mm on a 100 mm VAS.
- Total: Total of all reporting groups
Arm/Group | PF-04531083 1000 mg | PF-04531083 2000 mg | Ibuprofen 400 mg | Placebo | Total
Number analyzed (Participants) | 22 | 23 | 22 | 23 | 90
Age Continuous [Mean (Standard Deviation); unit: years] | 22.9 (3.7) | 23.4 (5.7) | 25.3 (4.5) | 25.3 (5.4) | 24.2 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 22 | 23 | 22 | 23 | 90

OUTCOME MEASURES:

1. Primary Outcome: Total Pain Relief (TOTPAR) Score From 0 to 6 Hours
Description: TOTPAR [6] was defined as the area under the pain relief (PR) curve through the first 6 hours after dosing. Area under the curve (AUC) was calculated using the trapezoid rule with PR was assumed to be 0 at time=0. PR assessed on a 5-point categorical scale; 0 (none), 1 (a little), 2 (some), 3 (a lot) and 4 (complete), at 15, 30, 45, minutes and at different time points during the study up to 6 hours post-dose. Total score range for TOTPAR [6]: 0 (worst) - 24 (best), higher value of TOTPAR indicated greater degree of PR.
Time Frame: 0 to 6 hours
Population: Full analysis set (FAS) included all randomized participants who had received at least 1 dose of study treatment and not received rescue medication of any type in the first 90 minutes following treatment administration. Missing PR values were imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: units on a scale*hour
Arm/Group | PF-04531083 1000 mg | PF-04531083 2000 mg | Ibuprofen 400 mg | Placebo
Number analyzed (Participants) | 22 | 23 | 22 | 23
units on a scale*hour | 4.3 (1.5) | 4.4 (1.5) | 8.8 (1.5) | 5.3 (1.5)
Statistical Analysis 1: Comparison: PF-04531083 1000 mg vs Placebo; Analysis of co-variance (ANCOVA) model was used with treatment as a fixed effect and baseline pain intensity as a covariate. LS mean estimates of the treatment difference along with 90 percent (%) confidence interval (CI) was presented; Test type: Superiority or Other; Least squares (LS) mean difference = -1.1, 90% CI 2-sided [-4.3 to 2.2], Standard Error of Mean 1.9
Statistical Analysis 2: Comparison: PF-04531083 2000 mg vs Placebo; ANCOVA model was used with treatment as a fixed effect and baseline pain intensity as a covariate. LS mean estimates of the treatment difference along with 90% CI was presented; Test type: Superiority or Other; LS mean difference = -0.9, 90% CI 2-sided [-4.1 to 2.3], Standard Error of Mean 1.9
Statistical Analysis 3: Comparison: Ibuprofen 400 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; LS mean difference = 3.5, 90% CI 2-sided [0.3 to 6.7], Standard Error of Mean 1.9

2. Secondary Outcome: Number of Participants With Peak Pain Relief (PPR)
Description: PPR was defined as the highest PR score achieved at any time point during the evaluation period, prior to rescue medication. PR was assessed on a 5-point categorical scale; 0 (none), 1 (a little), 2 (some), 3 (a lot) and 4 (complete).
Time Frame: 0 to 24 hours
Population: FAS included all randomized participants who had received at least 1 dose of study treatment and not received rescue medication of any type in the first 90 minutes following treatment administration.
Measure: Number; unit: participants
Arm/Group | PF-04531083 1000 mg | PF-04531083 2000 mg | Ibuprofen 400 mg | Placebo
Number analyzed (Participants) | 22 | 23 | 22 | 23
participants
  None | 4 | 3 | 3 | 4
  A Little | 4 | 6 | 3 | 4
  Some | 4 | 7 | 3 | 4
  A Lot | 5 | 0 | 6 | 5
  Complete | 5 | 7 | 7 | 6

3. Secondary Outcome: Time-specific Pain Relief (PR) Score
Description: PR was assessed on a 5-point categorical scale; 0 (none), 1 (a little), 2 (some), 3 (a lot) and 4 (complete) at each relevant time points.
Time Frame: 0, 15, 30, 45 minutes, 1, 1.5, 2, 3, 4, 6, 8, 24 hours, prior to rescue medication (RM)
Population: FAS included all randomized participants who had received at least 1 dose of study treatment and not received rescue medication of any type in the first 90 minutes following treatment administration. n=number of participants evaluable for this measure at specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-04531083 1000 mg | PF-04531083 2000 mg | Ibuprofen 400 mg | Placebo
Number analyzed (Participants) | 22 | 23 | 22 | 23
units on a scale
  0 hours (n=22, 23, 22, 23) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  15 minutes (n=22, 23, 22, 23) | 0.59 (0.80) | 0.78 (0.95) | 0.59 (0.91) | 0.57 (0.73)
  30 minutes (n=22, 23, 22, 23) | 0.82 (0.85) | 1.04 (1.07) | 1.23 (1.23) | 1.04 (1.02)
  45 minutes (n=22, 23, 22, 23) | 0.91 (0.87) | 1.26 (1.18) | 1.55 (1.22) | 1.35 (1.07)
  1 hour (n=22, 23, 22, 23) | 0.86 (0.99) | 1.13 (1.06) | 1.73 (1.28) | 1.39 (1.34)
  1.5 hours (n=22, 23, 22, 23) | 0.82 (0.91) | 0.91 (1.12) | 1.77 (1.38) | 1.30 (1.22)
  2 hours (n=15, 13, 20, 16) | 1.07 (0.96) | 1.77 (0.93) | 1.90 (1.37) | 1.63 (1.26)
  3 hours (n=11, 10, 15, 12) | 2.27 (0.79) | 2.30 (1.06) | 2.73 (0.96) | 2.25 (1.06)
  4 hours (n=11, 10, 15, 10) | 2.27 (0.79) | 2.20 (0.92) | 2.87 (0.92) | 2.60 (1.17)
  6 hours (n=11, 9, 15, 9) | 2.64 (0.67) | 2.67 (0.87) | 2.87 (0.92) | 3.11 (0.78)
  8 hours (n=10, 9, 15, 8) | 2.70 (0.82) | 2.67 (1.32) | 2.60 (0.91) | 3.13 (0.83)
  24 hours (n=8, 7, 8, 7) | 3.63 (0.52) | 3.86 (0.38) | 3.38 (0.74) | 3.71 (0.49)
  Prior to RM (n=14, 16, 14, 16) | 0.14 (0.36) | 0.25 (0.58) | 0.50 (0.65) | 0.25 (0.45)

4. Secondary Outcome: Time-specific Pain Intensity Difference (PID) Score
Description: Pain intensity was assessed on a categorical scale ranging from 0 (none), 1 (mild), 2 (moderate) and 3 (severe). PID was calculated as pain intensity at baseline minus pain intensity at the respective post-baseline visit.
Time Frame: 15, 30, 45 minutes, 1, 1.5, 2, 3, 4, 6, 8, 24 hours, prior to RM
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-04531083 1000 mg | PF-04531083 2000 mg | Ibuprofen 400 mg | Placebo
Number analyzed (Participants) | 22 | 23 | 22 | 23
units on a scale
  15 minutes (n=22, 23, 22, 23) | 0.14 (0.64) | 0.17 (0.65) | 0.18 (0.39) | 0.17 (0.39)
  30 minutes (n=22, 23, 22, 23) | 0.18 (0.73) | 0.35 (0.78) | 0.41 (0.67) | 0.35 (0.71)
  45 minutes (n=22, 23, 22, 23) | 0.23 (0.69) | 0.30 (0.88) | 0.59 (0.67) | 0.35 (0.83)
  1 hour (n=22, 23, 22, 23) | 0.14 (0.64) | 0.17 (0.83) | 0.68 (0.72) | 0.39 (1.03)
  1.5 hours (n=22, 23, 22, 23) | 0.00 (0.69) | 0.04 (0.88) | 0.68 (0.78) | 0.26 (1.01)
  2 hours (n=15, 13, 20, 16) | 0.13 (0.64) | 0.69 (0.48) | 0.75 (0.97) | 0.44 (0.96)
  3 hours (n=11, 10, 15, 12) | 0.82 (0.40) | 1.00 (0.67) | 1.20 (0.68) | 0.83 (0.94)
  4 hours (n=11, 10, 15, 10) | 0.91 (0.30) | 0.90 (0.57) | 1.20 (0.56) | 1.20 (0.63)
  6 hours (n=11, 9, 15, 9) | 0.91 (0.30) | 1.22 (0.44) | 1.20 (0.68) | 1.44 (0.53)
  8 hours (n=10, 9, 15, 8) | 1.00 (0.47) | 1.22 (0.67) | 1.20 (0.56) | 1.50 (0.76)
  24 hours (n=8, 7, 8, 7) | 1.63 (0.52) | 1.86 (0.38) | 1.63 (0.74) | 1.86 (0.69)
  Prior to RM (n=14, 16, 14, 16) | -0.57 (0.51) | -0.44 (0.51) | -0.29 (0.61) | -0.50 (0.52)

5. Secondary Outcome: Summed Pain Intensity Difference (SPID) Score at 6 Hours and 24 Hours
Description: Pain intensity was assessed on a categorical scale ranging from 0 (none), 1 (mild), 2 (moderate) and 3 (severe). PID was calculated as pain intensity at baseline minus pain intensity at the respective post-baseline visit. The SPID at 6 and 24 hours was derived by calculating the area under the PID effect curve through the first 6 or 24 hours post-dose respectively. The AUC was calculated using the trapezoid rule. Total score range: -6 (worst) to 18 (best) for SPID 0-6, and -24 (worst) to 72 (best) for SPID 0-24. Higher value of SPID indicated greater degree of pain relief.
Time Frame: 0 to 6, 0 to 24 hours
Population: FAS included all randomized participants who had received at least 1 dose of study treatment and not received rescue medication of any type in the first 90 minutes following treatment administration. Missing SPID values were imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: units on a scale*hour
Arm/Group | PF-04531083 1000 mg | PF-04531083 2000 mg | Ibuprofen 400 mg | Placebo
Number analyzed (Participants) | 22 | 23 | 22 | 23
units on a scale*hour
  SPID 0-6 | 0.9 (1.1) | 1.0 (1.1) | 4.1 (1.1) | 1.4 (1.1)
  SPID 0-24 | 4.7 (5.4) | 5.6 (5.3) | 13.3 (5.4) | 5.7 (5.3)
Statistical Analysis 1: Comparison: PF-04531083 1000 mg vs Placebo; SPID 0-6: LS mean estimates of the treatment difference along with 90% CI were based on ANCOVA model including treatment as a fixed effect and baseline pain intensity as a covariate; Test type: Superiority or Other; LS mean difference = -0.4, 90% CI 2-sided [-2.8 to 1.9], Standard Error of Mean 1.4
Statistical Analysis 2: Comparison: PF-04531083 2000 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; LS mean difference = -0.3, 90% CI 2-sided [-2.7 to 2.0], Standard Error of Mean 1.4
Statistical Analysis 3: Comparison: Ibuprofen 400 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; LS mean difference = 2.8, 90% CI 2-sided [0.4 to 5.1], Standard Error of Mean 1.4
Statistical Analysis 4: Comparison: PF-04531083 1000 mg vs Placebo; SPID 0-24: LS mean estimates of the treatment difference along with 90% CI were based on ANCOVA model including treatment as a fixed effect and baseline pain intensity as a covariate; Test type: Superiority or Other; LS mean difference = -1.0, 90% CI 2-sided [-12.6 to 10.5], Standard Error of Mean 7.0
Statistical Analysis 5: Comparison: PF-04531083 2000 mg vs Placebo; [analysis description as in outcome 5, analysis 4]; Test type: Superiority or Other; LS mean difference = -0.1, 90% CI 2-sided [-11.5 to 11.4], Standard Error of Mean 6.9
Statistical Analysis 6: Comparison: Ibuprofen 400 mg vs Placebo; [analysis description as in outcome 5, analysis 4]; Test type: Superiority or Other; LS mean difference = 7.6, 90% CI 2-sided [-4.0 to 19.1], Standard Error of Mean 7.0

6. Secondary Outcome: Total Pain Relief (TOTPAR) Score From 0 to 24 Hours
Description: TOTPAR [24] was defined as the area under the pain relief (PR) curve through the 24 hours after dosing. Area under the curve (AUC) was calculated using the trapezoid rule with PR assumed to be 0 at time=0. PR was assessed on a 5-point categorical scale; 0 (none), 1 (a little), 2 (some), 3 (a lot) and 4 (complete), at 15, 30, 45, minutes and at different time points during the study up to 24 hours post-dose. Total score range for TOTPAR [24]: 0 (worst) - 96 (best), higher value of TOTPAR indicated greater degree of PR.
Time Frame: 0 to 24 hours
Population: FAS included all randomized participants who had received at least 1 dose of study treatment and not received rescue medication of any type in the first 90 minutes following treatment administration. Missing TOTPAR values were imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: units on a scale*hour
Arm/Group | PF-04531083 1000 mg | PF-04531083 2000 mg | Ibuprofen 400 mg | Placebo
Number analyzed (Participants) | 22 | 23 | 22 | 23
units on a scale*hour | 21.8 (7.4) | 20.7 (7.3) | 30.8 (7.4) | 21.5 (7.3)
Statistical Analysis 1: Comparison: PF-04531083 1000 mg vs Placebo; LS mean estimates of the treatment difference along with 90% CI were based on ANCOVA model including treatment as a fixed effect and baseline pain intensity as a covariate; Test type: Superiority or Other; LS mean difference = 0.2, 90% CI 2-sided [-15.6 to 16.1], Standard Error of Mean 9.5
Statistical Analysis 2: Comparison: PF-04531083 2000 mg vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; LS mean difference = -0.8, 90% CI 2-sided [-16.5 to 14.8], Standard Error of Mean 9.4
Statistical Analysis 3: Comparison: Ibuprofen 400 mg vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; LS mean difference = 9.3, 90% CI 2-sided [-6.6 to 25.1], Standard Error of Mean 9.5

7. Secondary Outcome: Time to Onset of First Perceptible Pain Relief (PR)
Description: Participants evaluated the time to first perceptible relief by stopping a stopwatch labeled 'first perceptible relief' at the moment they first began to experience any relief.
Time Frame: 0 to 24 hours
Population: as for outcome 2
Measure: Median (90% Confidence Interval); unit: hours
Arm/Group | PF-04531083 1000 mg | PF-04531083 2000 mg | Ibuprofen 400 mg | Placebo
Number analyzed (Participants) | 22 | 23 | 22 | 23
hours | 0.4 [0.2 to 0.8] | 0.3 [0.2 to 0.4] | 0.4 [0.3 to 0.5] | 0.4 [0.3 to 0.5]
Statistical Analysis 1: Comparison: PF-04531083 1000 mg vs Placebo; Hazard Ratio (HR) estimates of the treatment difference along with 90% CI were based Cox proportional hazards model including treatment and baseline pain intensity as fixed effects; Test type: Superiority or Other; Hazard Ratio (HR) = 0.8, 90% CI 2-sided [0.5 to 1.5]
Statistical Analysis 2: Comparison: PF-04531083 2000 mg vs Placebo; HR estimates of the treatment difference along with 90% CI were based Cox proportional hazards model including treatment and baseline pain intensity as fixed effects; Test type: Superiority or Other; Hazard Ratio (HR) = 1.2, 90% CI 2-sided [0.7 to 2.1]
Statistical Analysis 3: Comparison: Ibuprofen 400 mg vs Placebo; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; Hazard Ratio (HR) = 1.1, 90% CI 2-sided [0.6 to 2.0]

8. Secondary Outcome: Time to Onset of First Meaningful Pain Relief (PR)
Description: Participants evaluated the time to first meaningful relief by stopping a second stopwatch labeled 'meaningful relief' at the moment they first began to experience meaningful relief.
Time Frame: 0 to 24 hours
Population: as for outcome 2
Measure: Median (90% Confidence Interval); unit: hours
Arm/Group | PF-04531083 1000 mg | PF-04531083 2000 mg | Ibuprofen 400 mg | Placebo
Number analyzed (Participants) | 22 | 23 | 22 | 23
hours | 3.0 [2.5 to 5.6] | 4.9 [2.0 to NA] — Upper limit of 90% confidence interval was not estimable due to empirical distribution of the data. | 3.3 [1.0 to 4.2] | 3.5 [2.8 to 4.1]
Statistical Analysis 1: Comparison: PF-04531083 1000 mg vs Placebo; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; Hazard Ratio (HR) = 1.0, 90% CI 2-sided [0.5 to 2.1]
Statistical Analysis 2: Comparison: PF-04531083 2000 mg vs Placebo; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; Hazard Ratio (HR) = 0.9, 90% CI 2-sided [0.4 to 1.8]
Statistical Analysis 3: Comparison: Ibuprofen 400 mg vs Placebo; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; Hazard Ratio (HR) = 1.5, 90% CI 2-sided [0.7 to 2.9]

9. Secondary Outcome: Time to First Use of Rescue Medication
Description: Time to first use of rescue medication (2 tablets of acetaminophen 500 mg as starting dose) was calculated by subtracting time of first administration of study medication from the rescue medication administration time.
Time Frame: 1.5 to 24 hours
Population: as for outcome 2
Measure: Median (90% Confidence Interval); unit: hours
Arm/Group | PF-04531083 1000 mg | PF-04531083 2000 mg | Ibuprofen 400 mg | Placebo
Number analyzed (Participants) | 22 | 23 | 22 | 23
hours | 4.8 [1.8 to NA] — Upper limit of 90% confidence interval was not estimable due to empirical distribution of the data. | 2.6 [1.7 to 10.4] | 11.1 [2.4 to NA] — Upper limit of 90% confidence interval was not estimable due to empirical distribution of the data. | 3.2 [2.0 to 12.9]
Statistical Analysis 1: Comparison: PF-04531083 1000 mg vs Placebo; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; Hazard Ratio (HR) = 1.0, 90% CI 2-sided [0.6 to 1.9]
Statistical Analysis 2: Comparison: PF-04531083 2000 mg vs Placebo; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; Hazard Ratio (HR) = 1.3, 90% CI 2-sided [0.7 to 2.4]
Statistical Analysis 3: Comparison: Ibuprofen 400 mg vs Placebo; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; Hazard Ratio (HR) = 0.7, 90% CI 2-sided [0.4 to 1.3]

10. Secondary Outcome: Number of Participants With Rescue Medication
Description: Participants who did not experience adequate pain relief after 90 minutes post-dose of study medication had received 2 tablets of acetaminophen 500 mg as rescue medication.
Time Frame: 0 to 24 hours
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | PF-04531083 1000 mg | PF-04531083 2000 mg | Ibuprofen 400 mg | Placebo
Number analyzed (Participants) | 22 | 23 | 22 | 23
participants | 14 | 16 | 14 | 16

11. Secondary Outcome: Participant Global Evaluation of Study Medication
Description: Participant rated the study medication that they received during the study, at both the 6 hour and 24 hour observations or at time of rescue medication, whichever occurs first, by answering the following question on 6-point categorical scale: how would you rate the study medication you received for pain? 5=excellent, 4=very good, 3=good, 2=fair and 1=poor.
Time Frame: 6, 24 hours, prior to RM
Population: FAS included all randomized participants who had received at least 1 dose of study treatment and not received rescue medication of any type in the first 90 minutes following treatment administration. Participants analyzed in this outcome for prior to rescue medication included only those participants who took rescue medication.
Measure: Number; unit: participants
Arm/Group | PF-04531083 1000 mg | PF-04531083 2000 mg | Ibuprofen 400 mg | Placebo
Number analyzed (Participants) | 22 | 23 | 22 | 23
participants
  6 hours: Excellent | 0 | 2 | 2 | 1
  6 hours: Very Good | 2 | 1 | 10 | 5
  6 hours: Good | 7 | 4 | 3 | 3
  6 hours: Fair | 1 | 2 | 0 | 0
  6 hours: Poor | 1 | 0 | 0 | 0
  6 hours: Not Done | 11 | 14 | 7 | 14
  24 hours: Excellent | 1 | 2 | 2 | 4
  24 hours: Very Good | 5 | 3 | 5 | 0
  24 hours: Good | 2 | 2 | 1 | 3
  24 hours: Fair | 0 | 0 | 0 | 0
  24 hours: Poor | 0 | 0 | 0 | 0
  24 hours: Not Done | 14 | 16 | 14 | 16
  Prior to RM: Excellent | 0 | 0 | 1 | 0
  Prior to RM: Very Good | 0 | 0 | 4 | 2
  Prior to RM: Good | 2 | 1 | 2 | 3
  Prior to RM: Fair | 4 | 4 | 2 | 2
  Prior to RM: Poor | 8 | 11 | 5 | 9

12. Secondary Outcome: Participant Satisfaction Questionnaire
Description: Participant's response to 2 questions about "how satisfied or dissatisfied they were with the study medication for PR and overall performance (OP)" was obtained on a 5 point categorical scale, 1=very dissatisfied, 2=somewhat dissatisfied, 3=neither satisfied nor dissatisfied, 4=somewhat satisfied and 5=very satisfied.
Time Frame: 6, 24 hours, prior to RM
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | PF-04531083 1000 mg | PF-04531083 2000 mg | Ibuprofen 400 mg | Placebo
Number analyzed (Participants) | 22 | 23 | 22 | 23
participants
  6 hours PR: Very Satisfied | 2 | 1 | 7 | 4
  6 hours PR: Somewhat Satisfied | 6 | 3 | 7 | 4
  6 hours PR: Neither Satisfied nor Dissatisfied | 1 | 3 | 1 | 1
  6 hours PR: Somewhat Dissatisfied | 2 | 2 | 0 | 0
  6 hours PR: Very Dissatisfied | 0 | 0 | 0 | 0
  6 hours PR: Not Done | 11 | 14 | 7 | 14
  6 hours OP: Very Satisfied | 3 | 2 | 5 | 5
  6 hours OP: Somewhat Satisfied | 6 | 4 | 9 | 3
  6 hours OP: Neither Satisfied nor Dissatisfied | 0 | 2 | 1 | 1
  6 hours OP: Somewhat Dissatisfied | 2 | 0 | 0 | 0
  6 hours OP: Very Dissatisfied | 0 | 1 | 0 | 0
  6 hours OP: Not Done | 11 | 14 | 7 | 14
  24 hours PR: Very Satisfied | 3 | 4 | 7 | 4
  24 hours PR: Somewhat Satisfied | 4 | 3 | 0 | 3
  24 hours PR: Neither Satisfied nor Dissatisfied | 1 | 0 | 1 | 0
  24 hours PR: Somewhat Dissatisfied | 0 | 0 | 0 | 0
  24 hours PR: Very Dissatisfied | 0 | 0 | 0 | 0
  24 hours PR: Not Done | 14 | 16 | 14 | 16
  24 hours OP: Very Satisfied | 3 | 2 | 7 | 4
  24 hours OP: Somewhat Satisfied | 4 | 5 | 0 | 3
  24 hours OP: Neither Satisfied nor Dissatisfied | 1 | 0 | 1 | 0
  24 hours OP: Somewhat Dissatisfied | 0 | 0 | 0 | 0
  24 hours OP: Very Dissatisfied | 0 | 0 | 0 | 0
  24 hours OP: Not Done | 14 | 16 | 14 | 16
  Prior to RM, PR: Very Satisfied | 0 | 0 | 5 | 0
  Prior to RM, PR: Somewhat Satisfied | 1 | 1 | 2 | 4
  Prior to RM, PR:Neither Satisfied nor Dissatisfied | 1 | 5 | 0 | 2
  Prior to RM, PR: Somewhat Dissatisfied | 4 | 2 | 2 | 3
  Prior to RM, PR: Very Dissatisfied | 8 | 8 | 5 | 7
  Prior to RM, OP: Very Satisfied | 0 | 0 | 3 | 0
  Prior to RM, OP: Somewhat Satisfied | 1 | 1 | 4 | 4
  Prior to RM, OP:Neither Satisfied nor Dissatisfied | 2 | 5 | 0 | 2
  Prior to RM, OP: Somewhat Dissatisfied | 3 | 2 | 1 | 3
  Prior to RM, OP: Very Dissatisfied | 8 | 8 | 6 | 7

13. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-04531083
Time Frame: 0 (pre-dose), 1, 2, 4, 6, 24 hours post-dose
Population: Pharmacokinetic (PK) analysis set included all randomized and treated participants for whom a PK sample was obtained and analyzed within the treatment period.
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-04531083 1000 mg | PF-04531083 2000 mg
Number analyzed (Participants) | 22 | 23
nanogram per milliliter (ng/mL) | 5761 (1905.0) | 9433 (3527.0)

14. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-04531083
Time Frame: 0 (pre-dose), 1, 2, 4, 6, 24 hours post-dose
Population: PK analysis set included all randomized and treated participants for whom a PK sample was obtained and analyzed within the treatment period.
Measure: Median (Full Range); unit: hours
Arm/Group | PF-04531083 1000 mg | PF-04531083 2000 mg
Number analyzed (Participants) | 22 | 23
hours | 4.02 [1.02 to 6.28] | 6.00 [2.02 to 24.2]

15. Secondary Outcome: Area Under the Curve From Time Zero to 6 Hour [AUC (0-6)] of PF-04531083
Description: AUC (0-6)= Area under the plasma concentration versus time curve from time zero (pre-dose) to 6 hours post-dose concentration.
Time Frame: 0 (pre-dose), 1, 2, 4, 6 hours post-dose
Population: as for outcome 14
Measure: Geometric Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | PF-04531083 1000 mg | PF-04531083 2000 mg
Number analyzed (Participants) | 22 | 23
nanogram*hour per milliliter (ng*hr/mL) | 21920 (7707.8) | 34640 (16408.0)

16. Secondary Outcome: Area Under the Curve From Time Zero to 24 Hour [AUC (0-24)] of PF-04531083
Description: AUC (0-24)= Area under the plasma concentration versus time curve from time zero (pre-dose) to 24 hours post-dose concentration.
Time Frame: 0 (pre-dose), 1, 2, 4, 6, 24 hours post-dose
Population: as for outcome 14
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | PF-04531083 1000 mg | PF-04531083 2000 mg
Number analyzed (Participants) | 22 | 23
ng*hr/mL | 80140 (23571) | 147100 (49215)

17. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Ibuprofen
Time Frame: 0 (pre-dose), 1, 2, 4, 6, 24 hours post-dose
Population: as for outcome 14
Measure: Geometric Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | Ibuprofen 400 mg
Number analyzed (Participants) | 22
microgram per milliliter (mcg/mL)
  (R)-Ibuprofen | 10.93 (4.6191)
  (S)-Ibuprofen | 12.10 (3.7848)

18. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Ibuprofen
Time Frame: 0 (pre-dose), 1, 2, 4, 6, 24 hours post-dose
Population: as for outcome 14
Measure: Median (Full Range); unit: hours
Arm/Group | Ibuprofen 400 mg
Number analyzed (Participants) | 22
hours
  (R)-Ibuprofen | 4.02 [1.00 to 24.1]
  (S)-Ibuprofen | 4.02 [1.02 to 6.23]

19. Secondary Outcome: Area Under the Curve From Time Zero to 6 Hour [AUC (0-6)] of Ibuprofen
Description: as for outcome 15
Time Frame: 0 (pre-dose), 1, 2, 4, 6 hours post-dose
Population: as for outcome 14
Measure: Geometric Mean (Standard Deviation); unit: microgram*hour per milliliter (mcg*h/mL)
Arm/Group | Ibuprofen 400 mg
Number analyzed (Participants) | 22
microgram*hour per milliliter (mcg*h/mL)
  (R)-Ibuprofen | 31.39 (12.847)
  (S)-Ibuprofen | 38.72 (13.070)

20. Secondary Outcome: Area Under the Curve From Time Zero to 24 Hour [AUC (0-24)] of Ibuprofen
Description: as for outcome 16
Time Frame: 0 (pre-dose), 1, 2, 4, 6, 24 hours post-dose
Population: as for outcome 14
Measure: Geometric Mean (Standard Deviation); unit: mcg*hr/mL
Arm/Group | Ibuprofen 400 mg
Number analyzed (Participants) | 22
mcg*hr/mL
  (R)-Ibuprofen | 56.82 (49.272)
  (S)-Ibuprofen | 82.58 (47.992)

21. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial/prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to Day 10 to 14.
Time Frame: Baseline up to Day 10-14 (Follow-up)
Population: Safety analysis set included all randomized participants who received at least 1 dose of study treatment.
Measure: Number; unit: participants
Arm/Group | PF-04531083 1000 mg | PF-04531083 2000 mg | Ibuprofen 400 mg | Placebo
Number analyzed (Participants) | 22 | 23 | 22 | 23
participants
  AEs | 13 | 12 | 11 | 9
  SAEs | 0 | 0 | 0 | 0

22. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Test Abnormality
Description: Hematology (hemoglobin, hematocrit, red blood cell count, platelets, leukocytes, total neutrophils, eosinophils, basophils, lymphocytes, monocytes); liver function (total bilirubin, direct bilirubin, indirect bilirubin, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, albumin, total protein); renal function (creatinine, blood urea nitrogen, uric acid, sodium, potassium, chloride, bicarbonate, calcium); urinalysis (urine pH, glucose, ketones, protein, blood, nitrite, leukocyte esterase), and clinical chemistry (glucose) were performed.
Time Frame: Baseline up to Day 10-14 (Follow-up)
Population: Safety analysis set included all randomized participants who received at least 1 dose of study treatment.
Measure: Number; unit: participants
Arm/Group | PF-04531083 1000 mg | PF-04531083 2000 mg | Ibuprofen 400 mg | Placebo
Number analyzed (Participants) | 22 | 23 | 22 | 23
participants | 4 | 6 | 5 | 6

23. Secondary Outcome: Supine Systolic and Diastolic Blood Pressure (BP)
Description: Supine systolic and diastolic BP was measured after the participant has been rested in the supine position for at least 5 minutes with the participant's arm supported at the level of the heart, and recorded to the nearest millimeters of mercury (mmHg). The same arm and position and same size BP cuff was used throughout the study.
Time Frame: Screening, Day 0, 1 (pre-dose), 2, 10-14 (Follow-up)
Population: Safety analysis set included all randomized participants who received at least 1 dose of study treatment. n=number of participants evaluable for this measure at specified time point.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | PF-04531083 1000 mg | PF-04531083 2000 mg | Ibuprofen 400 mg | Placebo
Number analyzed (Participants) | 22 | 23 | 22 | 23
mmHg
  Screening: Systolic BP (n=22, 23, 22, 23) | 124.3 (9.70) | 123.2 (9.62) | 122.4 (10.05) | 126.5 (10.22)
  Screening: Diastolic BP (n=22, 23, 22, 23) | 71.4 (8.75) | 69.7 (6.33) | 71.4 (6.99) | 72.8 (8.31)
  Day 0: Systolic BP (n=22, 23, 22, 23) | 128.2 (14.41) | 122.4 (10.14) | 126.7 (11.15) | 128.0 (10.80)
  Day 0: Diastolic BP (n=22, 23, 22, 23) | 71.8 (10.52) | 71.1 (6.68) | 71.6 (6.75) | 71.3 (9.10)
  Day 1: Systolic BP (n=22, 23, 22, 23) | 122.8 (12.69) | 126.8 (13.17) | 126.6 (14.40) | 124.1 (14.39)
  Day 1: Diastolic BP (n=22, 23, 22, 23) | 67.2 (8.89) | 71.1 (9.59) | 72.5 (9.61) | 70.7 (11.51)
  Day 2: Systolic BP (n=22, 23, 22, 23) | 121.2 (10.51) | 119.3 (10.52) | 124.0 (11.39) | 122.2 (12.31)
  Day 2: Diastolic BP (n=22, 23, 22, 23) | 65.9 (9.26) | 66.3 (7.07) | 67.7 (8.90) | 69.6 (8.48)
  Day 10-14 (Follow-up): Systolic BP(n=21,23,22,22 ) | 122.8 (11.05) | 124.9 (10.70) | 125.4 (11.14) | 122.5 (10.18)
  Day 10-14 (Follow-up): Diastolic BP(n=21,23,22,22) | 69.7 (11.32) | 70.6 (9.66) | 72.1 (5.56) | 72.3 (9.83)

24. Secondary Outcome: 12-Lead Electrocardiogram (ECG) Parameters (PR, QRS, QT, QTcF Intervals)
Description: Standard 12-lead ECG was performed after the participant has rested quietly for at least 10 minutes in a supine position. ECG intervals included PR interval (time between the onset of atrial depolarization and the onset of ventricular depolarization), QRS interval (represented ventricular depolarization) and QT interval (time corresponding to the beginning of depolarization to repolarization of the ventricles) corrected using Fridericia's formula (QTcF = QT divided by cube root of RR interval).
Time Frame: Screening, Day 1, 2, 10-14 (Follow-up)
Population: Safety analysis set included all randomized participants who received at least 1 dose of study treatment. n=number of participants evaluable for this measure at specified time points for each arm group respectively.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | PF-04531083 1000 mg | PF-04531083 2000 mg | Ibuprofen 400 mg | Placebo
Number analyzed (Participants) | 22 | 23 | 22 | 23
milliseconds
  Screening: PR Interval (n=22, 23, 22, 23) | 157.1 (27.69) | 156.0 (20.64) | 150.7 (23.17) | 156.4 (22.12)
  Screening: QRS Interval (n=22, 23, 22, 23) | 90.3 (8.33) | 95.8 (9.96) | 93.2 (8.74) | 93.7 (8.68)
  Screening: QT Interval (n=22, 23, 22, 23) | 398.4 (34.27) | 413.2 (34.29) | 410.7 (25.43) | 410.3 (26.56)
  Screening: QTcF Interval (n=22, 23, 22, 23) | 399.8 (16.34) | 403.6 (18.33) | 400.9 (16.33) | 404.0 (17.03)
  Day 1: PR Interval (n=22, 23, 22, 23) | 154.2 (21.51) | 148.7 (18.71) | 148.4 (23.81) | 152.5 (14.93)
  Day 1: QRS Interval (n=22, 23, 22, 23) | 89.7 (7.15) | 95.0 (9.96) | 91.5 (7.90) | 90.8 (8.96)
  Day 1: QT Interval (n=22, 23, 22, 23) | 372.0 (18.27) | 391.1 (27.39) | 388.7 (28.41) | 388.9 (28.00)
  Day 1: QTcF Interval (n=22, 23, 22, 23) | 388.5 (15.48) | 393.4 (18.82) | 395.3 (17.66) | 398.7 (15.14)
  Day 2: PR Interval (n=22, 23, 22, 23) | 156.9 (22.83) | 149.1 (17.79) | 150.8 (22.86) | 153.9 (18.33)
  Day 2: QRS Interval (n=22, 23, 22, 23) | 87.6 (7.63) | 93.7 (8.10) | 88.5 (11.73) | 90.4 (8.38)
  Day 2: QT Interval (n=22, 23, 22, 23) | 381.1 (24.91) | 395.5 (32.99) | 385.8 (32.91) | 396.7 (26.22)
  Day 2: QTcF Interval (n=22, 23, 22, 23) | 394.0 (14.76) | 397.9 (18.87) | 396.6 (19.03) | 404.2 (16.82)
  Day 10-14 (Follow-up): PR Interval (n=0, 0, 0, 1) | NA (NA) — As planned follow-up visit ECG was not done since no significant change was observed during the 6 and 24 hours post-dose ECGs. | NA (NA) — As planned follow-up visit ECG was not done since no significant change was observed during the 6 and 24 hours post-dose ECGs. | NA (NA) — As planned follow-up visit ECG was not done since no significant change was observed during the 6 and 24 hours post-dose ECGs. | 148.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Day 10-14 (Follow-up): QRS Interval (n=0, 0, 0, 1) | NA (NA) — As planned follow-up visit ECG was not done since no significant change was observed during the 6 and 24 hours post-dose ECGs. | NA (NA) — As planned follow-up visit ECG was not done since no significant change was observed during the 6 and 24 hours post-dose ECGs. | NA (NA) — As planned follow-up visit ECG was not done since no significant change was observed during the 6 and 24 hours post-dose ECGs. | 102.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Day 10-14 (Follow-up): QT Interval (n=0, 0, 0, 1) | NA (NA) — As planned follow-up visit ECG was not done since no significant change was observed during the 6 and 24 hours post-dose ECGs. | NA (NA) — As planned follow-up visit ECG was not done since no significant change was observed during the 6 and 24 hours post-dose ECGs. | NA (NA) — As planned follow-up visit ECG was not done since no significant change was observed during the 6 and 24 hours post-dose ECGs. | 360.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Day 10-14 (Follow-up): QTcF Interval(n=0, 0, 0, 1) | NA (NA) — As planned follow-up visit ECG was not done since no significant change was observed during the 6 and 24 hours post-dose ECGs. | NA (NA) — As planned follow-up visit ECG was not done since no significant change was observed during the 6 and 24 hours post-dose ECGs. | NA (NA) — As planned follow-up visit ECG was not done since no significant change was observed during the 6 and 24 hours post-dose ECGs. | 401.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.

25. Secondary Outcome: 12-Lead Electrocardiogram (ECG) Parameter (Heart Rate)
Description: Standard 12-lead ECG was performed after the participant has rested quietly for at least 10 minutes in a supine position. The time interval between consecutive heart beats (RR interval) was used to calculate heart rate.
Time Frame: Screening, Day 1, 2, 10-14 (Follow-up)
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | PF-04531083 1000 mg | PF-04531083 2000 mg | Ibuprofen 400 mg | Placebo
Number analyzed (Participants) | 22 | 23 | 22 | 23
beats per minute
  Screening (n=22, 23, 22, 23) | 62.2 (11.99) | 57.1 (10.02) | 56.5 (8.05) | 58.0 (8.54)
  Day 1 (n=22, 23, 22, 23) | 69.1 (10.30) | 61.7 (7.08) | 64.0 (9.51) | 65.8 (10.89)
  Day 2 (n=22, 23, 22, 23) | 67.2 (9.83) | 62.5 (11.60) | 66.3 (10.09) | 64.3 (8.26)
  Day 10-14 (Follow-up) (n=0, 0, 0, 1) | NA (NA) — As planned follow-up visit ECG was not done since no significant change was observed during the 6 and 24 hours post-dose ECGs. | NA (NA) — As planned follow-up visit ECG was not done since no significant change was observed during the 6 and 24 hours post-dose ECGs. | NA (NA) — As planned follow-up visit ECG was not done since no significant change was observed during the 6 and 24 hours post-dose ECGs. | 83.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.

26. Secondary Outcome: Supine Pulse Rate
Description: Supine pulse rate was measured in the brachial/radial artery for at least 30 seconds.
Time Frame: Screening, Day 0, 1 (pre-dose), 2, 10-14 (Follow-up)
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | PF-04531083 1000 mg | PF-04531083 2000 mg | Ibuprofen 400 mg | Placebo
Number analyzed (Participants) | 22 | 23 | 22 | 23
beats per minute
  Screening (n=22, 23, 22, 23) | 60.1 (13.08) | 56.2 (10.48) | 55.1 (7.97) | 57.0 (10.45)
  Day 0 (n=22,23,22,23) | 61.6 (8.56) | 61.3 (9.89) | 62.1 (10.23) | 63.1 (12.40)
  Day 1 (n=22,23,22,23) | 66.4 (10.06) | 59.5 (8.81) | 61.2 (7.32) | 59.4 (9.48)
  Day 2 (n=22,23,22,23) | 64.1 (9.59) | 60.6 (12.03) | 65.9 (8.71) | 62.7 (8.55)
  Day 10-14 (Follow-up) (n=21, 23, 22, 22) | 61.3 (9.91) | 60.4 (10.60) | 59.6 (11.81) | 62.0 (8.91)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | PF-04531083 1000 mg | PF-04531083 2000 mg | Ibuprofen 400 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/23 | 0/22 | 0/23
Other Adverse Events (participants affected / at risk) | 13/22 | 10/23 | 8/22 | 5/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04531083 1000 mg (N=22) | PF-04531083 2000 mg (N=23) | Ibuprofen 400 mg (N=22) | Placebo (N=23)
Nausea (Gastrointestinal disorders) | 4 | 3 | 3 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Tooth infection (Infections and infestations) | 3 | 0 | 2 | 1
Blood bilirubin increased (Investigations) | 0 | 2 | 0 | 0
Blood bilirubin unconjugated increased (Investigations) | 0 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 5 | 8 | 1 | 0
Headache (Nervous system disorders) | 6 | 4 | 1 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0

LIMITATIONS AND CAVEATS:
Study was terminated for futility based on results of interim analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.